CLINICAL TRIAL: NCT03038347
Title: Evaluation of an Internet-based Training Program to Improve Cross-cultural Competencies in Psychotherapists
Brief Title: Training of Cross-cultural Competencies in Psychotherapists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Cornelia Weise, Assistant Professor, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Cross-cultural psychotherapy
Record Dates: First submitted 2017-01-17; First posted 2017-01-31 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: cross-cultural competencies; internet-based training; cognitive-behavioural therapy (CBT); psychotherapy training; competence training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training (Experimental): In the training group, participants work six weeks on the training program, one module per week. The modules contain PDF-files with text-based information, video files, case studies with associated questions as well as practical exercises that participants perform independently. The main purpose of this intervention is the improvement of cross-cultural competencies in psychotherapists
  Interventions: Behavioral: Training
- Education only (Active Comparator): In the education only group, participants work six weeks on a slimmed down version of the training program. The modules only contain text-based information without any exercises. After completion, participants receive access to the practical exercises, case studies and video files as well. Main purpose of the education only group is to determine whether the practical part of the training program can offer additional benefit.
  Interventions: Behavioral: Education only
- Waiting control (No Intervention): Initially, participants do not receive any training contents. After a six week waiting period, they can participate in the training program as well. Modules are equivalent to those of the training group. Purpose of this group is to determine whether the training program is effective.

INTERVENTIONS:
Behavioral: Training — Six modules containing PDF-files with text-based information, video files, case studies with associated questions and practical exercises. Participants can download the modules and associated materials from an online platform they need to register for. They receive access to modules and associated exercises once a week. After six weeks the training is completed.
  Arms: Training
Behavioral: Education only — Six modules containing only PDF-files with text-based information. Participants can download the modules and associated materials from an online platform they need to register for. They receive access to modules once a week. After six weeks the education is completed.
  Arms: Education only

SUMMARY:
The purpose of this study is to determine whether a web-based training program with text-based information as well as practical exercises can improve cross-cultural competencies in therapists.

DETAILED DESCRIPTION:
As the number of patients from diverse cultures increases in psychotherapeutic care, cross-cultural competencies of therapists become increasingly important. In particular, mental health care of patients with immigration background needs to be improved as studies show that these patients drop out of treatment more often and benefit less from therapy. In addition, patients with immigration background and refugees show higher prevalences in mental illnesses. Nevertheless, evaluated training programs to improve cross-cultural competencies in psychotherapists are lacking. In particular, web-based training programs, which allow therapists to work time-flexible and at their own pace on a training, are, to date, missing completely.

For the current study, a web-based training program to improve therapists' cross-cultural competencies was developed. It is based on existing conceptions of cross-cultural competencies. The developed program consists of six modules with the following contents: definitions and conceptions of culture, the role of cross-cultural competencies in psychotherapy, the influence of prejudices and discrimination as well as the role of migration and acculturation, and culturally sensitive diagnostics. The modules contain PDF-files with text-based information, video files, case studies with associated questions as well as practical exercises. The main focus of the training is the participants' self-reflection concerning their conceptions of (their own) culture and their beliefs about culturally diverse patients. The training group will be compared to two other groups, i.e. an education only and a waitlist control group. Whereas the waitlist control group will not receive any training materials, the education only group will receive a slimmed down version of the training consisting only of text-based information files.

ELIGIBILITY:
Inclusion Criteria:

* current psychotherapeutic work
* Internet access
* sufficient German language skills
* ongoing or completed training in Psychotherapy

Exclusion Criteria:

* too much previous knowledge about cross-cultural competencies (> 10h training)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Transcultural Competencies of Psychotherapists Questionnaire (TKKP; Reichardt et. al., in prep.) | pre-training, post-training (6 weeks after the start of the training); follow up (6 month after training completion)
  Change in cross-cultural psychotherapeutic competencies
Multicultural Counseling Inventory (MCI; Sodowsky, 1994) | pre-training, post-training (6 weeks after the start of the training); follow-up (6 month after training completion)
  Change in cross-cultural psychotherapeutic competencies

SECONDARY OUTCOMES:
Cultural sensitivity in actual psychotherapeutic work I | pre-training, post-training (6 weeks after the start of the training), follow-up (6 month after training completion)
  Percentage of culturally diverse patients currently in treatment in own actual psychotherapeutic work
Cultural sensitivity in actual psychotherapeutic work II | pre-training, post-training (6 weeks after the start of the training), follow-up (6 month after training completion)
  Willingness to treat culturally diverse patients in own actual psychotherapeutic work (rating scale)
Cultural sensitivity in actual psychotherapeutic work III | pre-training, post-training (6 weeks after the start of the training), follow-up (6 month after training completion)
  Satisfaction with cross-cultural therapies provided in actual psychotherapeutic work (rating scale)
Cultural sensitivity in actual psychotherapeutic work IV | pre-training, post-training (6 weeks after the start of the training), follow-up (6 month after training completion)
  Perceived competence in the currently provided cross-cultural therapies (rating scale)
Knowledge regarding the provision of cross-cultural psychotherapy | post-training (6 weeks after the start of the training)
  Test of specific knowledge gained during the training (knowledge test in multiple choice answer format)
Training satisfaction scale | post-training (6 weeks after the start of the training); follow-up (6 month after training completion)
  Satisfaction with the training (rating scale; items assessing satisfaction with contents and structure of the developed training)
Learning success scale | post-training (6 weeks after the start of the training); follow-up (6 month after training completion)
  Rating of competencies achieved through the training for the treatment of culturally diverse patients (rating scale, rating of the degree to which certain competencies have been achieved)
Cultural sensitivity in psychotherapeutic work (Behavioural change measure) | post-training (6 weeks after the start of the training), 2 months after training completion; follow-up (6 month after training completion)
  Rating of different case examples with focus on expected difficulty and effectiveness of psychotherapy (given different cases with different disorders, severity levels, and cultural backgrounds)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Weise, PhD, Principal Investigator — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg; Winfried Rief, PhD, Study Chair — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg; Ulrike von Lersner, PhD, Study Chair — Department of Transcultural Psychology, Humboldt University Berlin; Gerhard Andersson, PhD, Study Chair — Department of Behavioural Sciences and Learning, Linköping University
Locations (1):
- Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazel M, Wheeler J, Danesh J. Prevalence of serious mental disorder in 7000 refugees resettled in western countries: a systematic review. Lancet. 2005 Apr 9-15;365(9467):1309-14. doi: 10.1016/S0140-6736(05)61027-6. PMID 15823380
- [Background] Gaitanides, S. (2001). Zugangsbarrieren von Migrant (inn) en zu den sozialen und psychosozialen Diensten und Strategien interkultureller Öffnung. In G. Auernheimer (Hrsg.), Migration als Herausforderung für pädagogische Institutionen (pp. 181-194). Wiesbaden: Springer Fachmedien.
- [Background] Mösko, M., Baschin, K., Längst, G., & von Lersner, U. (2012). Interkulturelle Trainings für die psychosoziale Versorgung. Psychotherapeut, 57(1), 15-21.
- [Background] Mosko MO, Pradel S, Schulz H. [The care of people with a migration background in psychosomatic rehabilitation]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2011 Apr;54(4):465-74. doi: 10.1007/s00103-011-1245-x. German. PMID 21465403
- [Background] Reichardt, J., von Lersner, U., Rief, W., & Weise, C. (in Vorb.). Entwicklung und Validierung des Inventars zur Erfassung transkultureller Kompetenzen bei Psychotherapeuten (TKKP).
- [Background] Sodowsky, G. R., Taffe, R. C., Gutkin, T. B., & Wise, S. L. (1994). Development of the Multicultural Counseling Inventory: A Self-Report Measure of Multicultural Competencies. Journal of Counseling Psychology, 41(2), 137-148.
- [Background] Sue, D. W., Arredondo, P., & McDavis, R. J. (1992). Multicultural counseling competencies and standards: A call to the profession. Journal of Counseling & Development, 70(4), 477-486.
- [Background] Reichardt, J., von Lersner, U., Rief, W., & Weise, C. (2017). Wie lassen sich transkulturelle Kompetenzen bei Psychotherapeuten steigern? Vorstellung eines webbasierten Trainingsprogramms [How to improve cross-cultural competencies in psychotherapists? Introduction of a web-based training program]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie, 65(3), 155-165. doi:10.1024/1661-4747/a000316